CLINICAL TRIAL: NCT07390084
Title: Exploring the Decision to Drink (More) Alcohol Following Manipulations of Stress and Social Context
Acronym: DoraR00
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jonas Dora, Acting Assistant Professor, University of Washington
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00023737; R00AA030591 (NIH)
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Psychological Stress; Social Interaction
Keywords: stress induction; value-based decision-making
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stress Alone (Experimental): These participants will undergo a stress induction and will make decisions about consuming alcohol alone.
  Interventions: Other: Stress
- Stress Social (Experimental): These participants will undergo a stress induction and will make decisions about consuming alcohol with a known peer.
  Interventions: Other: Stress; Other: Social Context
- Control Alone (Experimental): These participants will undergo a control induction and will make decisions about consuming alcohol alone.
  Interventions: Other: Stress; Other: Social Context
- Control Social (Experimental): These participants will undergo a control induction and will make decisions about consuming alcohol with a known peer.
  Interventions: Other: Social Context

INTERVENTIONS:
Other: Stress — Participants randomly assigned to the stress condition will undergo the standard protocol of the Trier Social Stress Test. Participants randomly assigned to the control condition will undergo a validated, non-stressful control procedure mirroring the TSST.
  Arms: Control Alone; Stress Alone; Stress Social
Other: Social Context — Participants randomly assigned to the social condition will make decisions about consuming alcohol with a known peer. Participants randomly assigned to the control condition will make decisions about consuming alcohol alone.
  Arms: Control Alone; Control Social; Stress Social

SUMMARY:
This preregistration documents an experiment examining the effects of acute stress and social context on alcohol-related decision-making. The study uses a 2x2 factorial design (stress vs. control × social vs. alone) with dyadic recruitment.

DETAILED DESCRIPTION:
Behavioral data:

Our first set of hypotheses tests whether the decision is influenced by stress and social context:

H1a: Stress affects the decision between alcoholic and non-alcoholic drinks, so that participants in the stress conditions choose alcoholic over non-alcoholic drinks more often compared to participants in the no stress conditions.

H1b: Social context affects the decision between alcoholic and non-alcoholic drinks, so that participants in the social conditions choose alcoholic over non-alcoholic drinks more often compared to participants in the alone conditions.

H1c: We test two competing predictions:

(I) The effect of stress on the decision between alcohol and non-alcoholic drinks is modulated by social context, so that the effect of stress is stronger for participants that are in the social condition.

(II) The effect of stress on the decision between alcohol and non-alcoholic drinks is modulated by social context, so that the effect of stress is weaker for participants that are in the social condition

Drift diffusion modeling:

Our second set of hypotheses test how the decision might be influenced by stress and social context:

H2a: Stress affects the bias (but not the drift rate or boundary) parameter of the drift diffusion model, so that the bias parameter is more positive for participants in the stress conditions.

H2b: Social context affects the bias (but not the drift rate or boundary) parameter of the drift diffusion model, so that the bias parameter is more positive for participants in the social conditions.

H2c: Stress and social context have an interactive effect on the bias (but not the drift rate or boundary) parameter of the drift diffusion model, so that the bias parameter is either more or less positive for stressed participants who are in the social condition (in line with H1c).

ELIGIBILITY:
Inclusion Criteria:

* Drinking alcohol at least once a week
* Consuming 4 (female) or 5 (male) drinks in one occasion at least once a month

Exclusion Criteria:

* Currently pregnant or trying to become pregnant
* Past or current treatment for alcohol use
* Past or current medical condition that contraindicates alcohol use
* Past or current reaction to alcohol that contraindicates alcohol use
* Past or current medication that contraindicates alcohol use

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of choices for alcoholic over non-alcoholic drinks. | 5 minutes
  Each participant will complete a two alternative forced-choice task in which they make repeated decisions between alcoholic and non-alcoholic drinks.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Dora, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data needed to reproduce our analyses will be shared on the Open Science Framework once the study has been completed.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Once data collection has been finalized and indefinitely.
Access Criteria: Everyone will be able to access the data, they will be public. All data we share are fully anonymized and not sensitive.
URL: https://osf.io/j9bkq/